CLINICAL TRIAL: NCT04534023
Title: A Randomized, Double-blind, Multi-center Clinical Study of the Efficacy of Idebenone in the Treatment of Primary Rapid Eye Movement Sleep Behavior Disorder Into Synucleinopathies
Brief Title: A Clinical Study of the Efficacy of Idebenone in the Treatment of iRBD Into Synucleinopathies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Second Affiliated Hospital of Soochow University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ruijinlj
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-11

CONDITIONS: Rapid Eye Movement Sleep Behavior Disorder; Synucleinopathy
MeSH Terms: conditions — REM Sleep Behavior Disorder; Synucleinopathies | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental): Idebenone
  Interventions: Drug: Idebenone
- control group (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Idebenone — trial group
  Arms: trial group
Drug: Placebo — control group
  Arms: control group

SUMMARY:
142 cases of patients with iRBD will be recruited from the neurology department of Ruijin Hospital, th second Affiliated Hospital of Soochow University and wuhan Union Hospital. After the informed consent was signed, they were divided into a trial group and a control group randomly. Each group contains 71 cases. The patients in the trial group will be treated with Idebenone, while the patients in the control group was treated with placebo. Both groups of subjects will be treated for 5 years, and patients will be followed-up and evaluated in the first year, 3 years and 5 years after treatment. The observations include the MDS-UPDRS questionnaires evaluation, blood biomarker measurements and fMRI or PET-MR examination to make sure whether the patients has converted to synucleinopathies. Study hypothesis: Idebenone therapy for patients with iRBD is safe and effective in delaying disease progression into synucleinopathies.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosed of iRBD.
2. Age between 40 and 75.
3. Be voluntarily to participate in the experiment by signing an informed consent form.

Exclusion Criteria:

1. Sleep apnea hypopnea syndrome
2. Slow movement, muscle rigidity, tremor or postural instability.
3. Neurological diseases such as cerebral hemorrhage, cerebral infarction, brain trauma, brain tumor or central nervous system infection.
4. Other sleep disorders or seizures.
5. Alcoholism or drug addiction patients.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Effective | 5 years
  5-year conversion rate of iRBD patients to synucleinopathies decreased
Ineffective | 5 years
  5-year conversion rate of iRBD patients to synucleinopathies remained unchanged or increased.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li Y, Wang C, Luo N, Chen F, Zhou L, Niu M, Kang W, Liu J. Efficacy of idebenone in the Treatment of iRBD into Synucleinopathies (EITRS): rationale, design, and methodology of a randomized, double-blind, multi-center clinical study. Front Neurol. 2022 Sep 12;13:981249. doi: 10.3389/fneur.2022.981249. eCollection 2022. PMID 36172027